CLINICAL TRIAL: NCT00771225
Title: A National Multicentric Randomised Study of the Correction of Genital Prolapse With Fascial Repair or Mesh (Prolift)
Brief Title: National,Multicentric Randomised Study of the Correction of Genital Prolapse With Fascial Repair or Mesh-Prolift
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: University of Sao Paulo General Hospital (Other); Irmandade da Santa Casa de Misericordia de Sao Paulo (Other); Federal University of São Paulo (Other); Feculdade de Medicina da Universidade de Sao Paulo - Brasil (Other)
Responsible Party: Johnson&Johnson, Hospital Universitario da Universidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 300-07-002
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2008-10

CONDITIONS: Genital Prolapse
Keywords: genital prolapse; surgery; fascial repair; mesh; prolift
MeSH Terms: interventions — Melanocyte-Stimulating Hormones

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- prolapse surgery with fascial repair (Other)
  Interventions: Procedure: fascial repair; Procedure: mesh repair
- prolapse surgery with mesh repair (Other)
  Interventions: Procedure: fascial repair; Procedure: mesh repair

INTERVENTIONS:
Procedure: fascial repair — surgery to treat genital prolapse with fascia repair
  Other Names: prolapse repair withouth mesh; prolapse repair with mesh; prolift
Procedure: mesh repair — surgery to genital prolapse with mesh
  Other Names: prolapse repair withouth mesh; prolapse repair with mesh; prolift

SUMMARY:
180 women with genital prolapse will be submitted to genital prolapse surgical correction, half of them with human fascia, and the other half with Prolift.

DETAILED DESCRIPTION:
180 women with genital prolapse will be submitted to genital prolapse surgical correction, half of them with human fascia, and the other half with Prolift.Are eligible women aged between 50 and 80 years old.

ELIGIBILITY:
Inclusion Criteria:

* Between 50 and 80 yrs

Exclusion Criteria:

* Less than 50 and more than 80 yrs

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2008-11; Primary Completion 2012-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Correction of genital prolapse | 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Simone Brandao, Principal Investigator — University of Sao Paulo
Locations (1):
- Simone Brandao, São Paulo, São Paulo, Brazil